CLINICAL TRIAL: NCT04422886
Title: Evaluating the Use of Transcranial Direct Current Stimulation as an Adjunct to Physiotherapy in Children and Youth With Acquired Brain Injury: Does Physiotherapy Plus Brain Stimulation Equal Better Motor Recovery?
Brief Title: Does Physiotherapy Plus Non-invasive Brain Stimulation Improve Motor Recovery in Children With Acquired Brain Injury?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low eligibility rate indicated that the study was not feasible
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-857
Record Dates: First submitted 2020-03-04; First posted 2020-06-09 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Acquired Brain Injury; Recovery of Function; Transcranial Electrical Stimulation
Keywords: physical therapy; pediatric; motor recovery; transcranial direct current stimulation
MeSH Terms: conditions — Brain Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: 2-arm parallel group feasibility randomized control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Physiotherapists providing treatment, physiotherapists conducting assessment, research coordinator, principal investigators, participants are all blinded to treatment allocation. Research assistants administered the transcranial direct current stimulation are not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Physio+tDCS (Experimental): Receives 20 minutes of active tDCS immediately prior to physiotherapy session, 4 days per week for a total of 16 sessions.
  Interventions: Device: active transcranial direct current stimulation (tDCS); Behavioral: Physiotherapy
- Physio+sham (Sham Comparator): Receives 20 minutes of sham tDCS immediately prior to physiotherapy session, 4 days per week for a total of 16 sessions.
  Interventions: Behavioral: Physiotherapy; Device: sham transcranial direct current stimulation (sham)

INTERVENTIONS:
Device: active transcranial direct current stimulation (tDCS) — 20 minutes at 2.0 mA with electrodes positioned at Cz and Fpz (as per 10-20 electrode placement guidelines)
  Arms: Physio+tDCS
Behavioral: Physiotherapy — motor skills based physiotherapy intervention (representative of typical goal-focused intervention in the clinical ABI program at Holland Bloorview), 45 minutes in duration
Device: sham transcranial direct current stimulation (sham) — 1 minutes at 1.0 mA with electrodes positioned at Cz and Fpz (as per 10-20 electrode placement guidelines) and 19 minutes with unit shut off and electrodes remaining on the scalp
  Arms: Physio+sham

SUMMARY:
The current study will evaluate the feasibility of transcranial direct current stimulation (tDCS) combined with an existing intensive physiotherapy program for children with ABI within the in/day-patient brain injury program at Holland Bloorview Kids Rehabilitation Hospital, Toronto, Canada. This feasibility randomized control trial will allocate 30 participants with ABI (age 5 to 18 years) to one of two treatment groups. One group will receive active tDCS prior to four of their existing physiotherapy sessions each week for a total of 16 sessions while the other group will receive sham/placebo tDCS prior to their physiotherapy sessions. Recovery of gross motor function will be compared between groups after the four weeks of tDCS treatment and again after three months to evaluate the short and longer-term impact of tDCS on an existing intensive physiotherapy program. Feasibility will be evaluated by tracking process, resource, and treatment indicators such as eligibility, enrollment, adherence, and tolerance rates.

DETAILED DESCRIPTION:
Objectives

The purpose of this study is to test the feasibility of using tDCS as a pre-treatment adjunct to intensive physiotherapy (the 'physio+tDCS' protocol) for children with ABI in the inpatient brain injury program at Holland Bloorview. The primary objectives of our study are to answer the following questions:

1. Is it feasible to implement a 'physio+tDCS' protocol within an existing inpatient ABI rehabilitation program based on participant eligibility, recruitment, tolerance, retention, and adherence to treatment protocol (e.g. session frequency and completion timelines)?
2. What is the effect of using tDCS as an adjunct to intensive physiotherapy on the recovery of gross motor function in children with moderate to severe ABI, as measured by individualized goal achievement and standardized gross motor outcome measures? METHODS Trial design Using a feasibility randomized control trial (RCT) study design, 30 children with moderate to severe ABI, enrolled in intensive brain injury rehabilitation at Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, will be randomized to the active or sham (control) tDCS intervention, which will be paired with individualized intensive physiotherapy (i.e., 'physio+tDCS' and 'physio+sham').

Randomization and Blinding Once enrolled in the study, an independent research assistant (RA) will randomly assign each child to the "sham" or "active" tDCS treatment group using a computer randomization web-based program and approach described below. Only the RAs involved in the study will be aware of each participant's treatment group assignment. The participants and the assessing/treating PTs will be blinded to the participant's treatment group.

Intervention tDCS Treatment- Depending on treatment group allocation, participants will receive 20 minutes of active tDCS or sham tDCS (provided by a trained RA) immediately prior to four of their physiotherapy sessions each week over 4 weeks for a total of 16 sessions. Children and PTs will be blinded to their tDCS/sham allocation. Two electrodes (5x7cm) in size will be used such that the anodal electrode will be attached to the Cz position on the scalp, to target the lower extremity region of bilateral primary motor cortices, and the cathodal electrode will be attached to the central supraorbital (Fpz) area of the forehead (20). Each tDCS treatment will consist of up to 2.0 mA of stimulation, adjusting for the child's age, head size, and tolerance as required. Participants will be told which treatment group they were allocated to after completing their final assessment (3 months after completing the treatment protocol). Participant symptoms and safety will be tracked before, during, and after each tDCS session. Adverse events reported via a REB-approved standard process to an independent in-house safety monitoring committee (SMC).

Physiotherapy Intervention- The physiotherapy treatment paired with the tDCS/sham consists of the typical motor skills-based physiotherapy children receive in the in/day-patient brain injury program at Holland Bloorview. Each 45- minute physiotherapy session promotes motor learning by focusing on functional tasks related to the child's personalized motor goals. Therapists individualize the program by adapting the tasks, instructions, feedback, and the level of challenge based on the child's needs.

Outcomes Feasibility- Feasibility of study implementation and tDCS will be evaluated by tracking process, resource, and treatment indicators. A priori feasibility targets are as follows: 20% of children admitted to the program will be eligible for the study, 70% of eligible children will be recruited; 80% of children will tolerate at least 1.0mA for 10 minutes of each tDCS session, 75% of treatment sessions will be completed, 95% of first reassessments will occur, and 80% of follow-up reassessments will occur at 3 months post-treatment. Adherence to the study protocol will be tracked by the number of tDCS and physiotherapy sessions scheduled per week and the number actually completed. Reasons for cancelled sessions or decreased number of sessions booked will be documented. Because tDCS should optimally occur in the half hour prior to physiotherapy, the start time and duration of stimulation will be documented, as well as the start time and duration of each physiotherapy session, on tracking sheets that will be completed by the RA/therapist conducting each tDCS/physiotherapy session. Eligibility data will be tracked across the study's duration to determine the proportion of children in the brain injury program who are eligible for the study, and the number who enrol and reasons for being excluded from the study will be documented.

Gross Motor- Baseline assessments will be conducted by a blinded independent PT assessor within four days of beginning the study treatment protocol. The first reassessment will be conducted by the same blinded PT assessor within four days after their last study intervention session. Three months after completion of the study treatment, a second reassessment will take place, involving the same outcome measures. Additional information regarding the participant's physiotherapy services (e.g., frequency, duration, focus of intervention) and amount of daily physical activity (e.g., frequency, duration, intensity, type) since study completion will also be recorded.

A priori targets for the co-primary gross motor outcomes are as follows: The active tDCS group should have at least 5 mean points of change more than the sham group on the Gross Motor Function Measure (GMFM) and at least 2.0 mean points of change more than the sham group on the Canadian Occupational Performance Measure (COPM).

ELIGIBILITY:
Inclusion Criteria:

* sustained a cerebral stroke (ischaemic or haemorrhage) or TBI within the last three months;
* admitted to Holland Bloorview for intensive brain injury rehabilitation in the in/day patient programs;
* medically stable, as determined by their primary physician at Holland Bloorview;
* receiving active motor learning-based physiotherapy intervention four to five times per week, as prescribed by their treating PT;
* tolerate approximately 45 minutes of physiotherapy intervention;
* able to sit at the edge of the bed independently for 5s
* capable of participating in standardized physiotherapy assessment, from a cognitive and behavioural perspective, and;
* able to communicate discomfort (verbally or non-verbally).

Exclusion Criteria:

* primary injury of the cerebellum
* pre-existing seizure disorder (i.e., prior to ABI);
* anti-seizure medication not optimized at the time of study enrollment (i.e., physician is actively adjusting type or dose of anti-seizure medication)
* brain tumour;
* metal implants in the head;
* cranial bone flap removed;
* stitches/staples or open wound on the head;
* experience with tDCS in the last two years (as knowledge of the sensation of active tDCS will affect blinding of treatment groups);
* diagnosed with another neurological disorder(s) affecting gross motor function (e.g., cerebral palsy, spinal cord injury, guillain-barre syndrome, etc…);
* requires more than 15 minutes per physiotherapy treatment session of non-motor learning content (e.g., behavioural redirection, craniosacral therapy, vestibular therapy, passive range of motion)
* lower extremity weight bearing activity restrictions secondary to injuries (e.g., fracture, ligamentous injury)(at the time of study enrollment)
* non-orthopaedic physical activity restrictions secondary to other injuries (e.g., splenic laceration)
* balances on most affected leg for greater than 5s
* enrolment in another treatment-based research study

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure | Change from baseline to 1st reassessment (4 weeks) to 2nd reassessment (3 months)
  A standardized physiotherapy assessment (validated for children with ABI) that assesses gross motor function in five dimensions (A- lying & rolling, B- sitting, C- crawling & kneeling, D- standing, walking, E-running & jumping). Each of the 88 items is scored from 0-3.
Canadian Occupational Performance Measure | Change from baseline to 1st reassessment (4 weeks) to 2nd reassessment (3 months)
  The Canadian Occupational Performance Measure is a standardized outcome measure that allows children and families to set goals and evaluate their performance and satisfaction with each goal on a scale of 1 to 10, where higher ratings mean increased performance and satisfaction. In this study, the goals will be participation-based goals related to gross motor activities.
Eligibility Rate | Through study completion, an average of two years
  The proportion of eligible participants compared to the number of children admitted for inpatient brain injury rehabilitation. Reported as a percentage.
Enrollment Rate | Through study completion, an average of two years
  The proportion of eligible participants who enrollment in the study. Reported as a percentage
Adherence Rate | Through study completion, an average of two years
  The proportion of enrolled participants who complete at least 12 of the 16 transcranial direct current stimulation (followed by physiotherapy) sessions.
Transcranial Direct Current Stimulation Tolerance | Through study completion, an average of two years
  The mean dose (measured in milliamperes) of transcranial direct current stimulation each participant receives.
Transcranial Direct Current Stimulation Tolerability Questionnaire | 1st reassessment (after 4-week treatment protocol)
  At baseline the participant indicate the most enjoyable and least enjoyable activity they have experienced in the last month. They order these two activities in relation to 7 familiar childhood experiences (e.g., watching TV, going to the dentist, going for a long car ride). At followup, the child is presented with the baseline ordering of these 9 activities and asked to indicate where transcranial direct current stimulation fits in the order (e.g. more enjoyable than going to the dentist but less enjoyable than watching TV).

SECONDARY OUTCOMES:
Acquired Brain Injury Challenge Assessment | Change from baseline to 1st reassessment (4 weeks) to 2nd reassessment (3 months)
  An 18-item standardized assessment of high level gross motor skills in children and youth with ABI. Each item assesses the child's ability to perform a skill and is scored on a 5-point scale according to time and quality of movement (where '5' indicates normal quality of movement and/or completion within a minimum amount of time while '0' indicates they were unable to complete the item within a maximum period of time and did not meet the criteria for quality).
10 metre fastest walk test | Change from baseline to 1st reassessment (4 weeks) to 2nd reassessment (3 months)
  Timed walk test over 10m with the participant walking as fast as possible.
Goal Attainment Scaling | Change from baseline to 1st reassessment (4 weeks) to 2nd reassessment (3 months)
  Participant-specific mobility, balance, and/or gross motor goals created by the treating physiotherapist to target specific activities they will work on in physiotherapy. The child's baseline ability is scored as a '-2'. The physiotherapist sets individualized targets for the child where '-1' indicates they are performing somewhat less than expected, '0' indicates they are performing at the expected level for a given time frame, '+1' indicates they have done somewhat better than expected, and '+2' indicates they have done much better than expected. When the goal is set, the physiotherapist sets '0' (the expected level) based on the timing of the reassessment and what they think the child is clinically capable of accomplishing in that time period.
Pediatric Evaluation of Disability Inventory (Mobility and Self-Care domains) | Change from baseline to 1st reassessment (4 weeks) to 2nd reassessment (3 months)
  Parent-reported computerized questionnaire evaluating their child's function ability. Each item is rated on 4-point scale where '0' indicates the child is unable to do and '4' indicates the activity is easy to do. A higher score indicates higher levels of independence with mobility and self-care.

CONTACTS AND LOCATIONS:
Overall Officials: Deryk S Beal, PhD, Principal Investigator — Clinician Scientist; Virginia Wright, PhD, Principal Investigator — Clinican Scientist
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
At this time data will not be shared with other researchers.